CLINICAL TRIAL: NCT03202290
Title: BANCO Study: Behavioral Addictions and Related NeuroCOgnitive Aspects: A Monocentric, Prospective, Controlled, Open-label Study of a Sample of Patients With Gambling Disorder
Acronym: BANCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC17_0165
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gambling disorder (Other): patients suffering from gambling disorder
  Interventions: Behavioral: Cognitive and clinical assessment
- Controls (Other): healthy controls
  Interventions: Behavioral: Cognitive and clinical assessment

INTERVENTIONS:
Behavioral: Cognitive and clinical assessment — The content of the assessment will be the same for all subjects and will consist of a cognitive assessment (neurocognition, social cognition, metacognition, emotional reactivity) and a clinical assessment (impulsivity, personality, psychriatric and addictive comorbidities)

SUMMARY:
The prevalence of people suffering from gambling disorder is relatively high, and the impact on this disorder the individual and those around him is considerable. The etiopathogenic model of gambling disorder is multifactorial, involving various risk and vulnerability factors, involved in the initiation and maintenance of the disorder. Among these factors, neurocognitive alterations associated with the disorder has recently aroused interest among researchers. In this study, the investigators propose to explore the neurocognitive impairments of patients suffering from gambling disorder compared to a control group, in order to identify alterations that could be the target of cognitive remediation programs. Gambling disorder provides a unique opportunity to study the specific neurocognitive impairments of the addictive process because it is not biased by the neurotoxic effect of substances as it is the case in substance use disorders.

ELIGIBILITY:
Inclusion Criteria:

* For the patients :

Aged of more than 18, Suffering from gambling disorder(diagnosis according to DSM-5), Patient starting care in the Addictology and Psychiatry department of the Nantes University Hospital, Mastering the French language, Social Security Affiliates, Having given consent

* For the volunteers:

Aged of more than 18, Subject not suffering from gambling disorder, Mastering the French language, Social Security Affiliates Having given consent

Exclusion Criteria:

* For patients :

Having psychiatric and addictive disorders (present and not stabilized mood disorders, anxiety disorders and substance-use disorders except nicotine, lifetime psychotic syndrome, diagnosed by the MINI and after consultation with the clinician), Unstable endocrine disruptions or neurological disorders (such as head trauma, neurodegenerative diseases, unbalanced epilepsy, mental retardation, etc.), Taking a non-stabilized psychotropic treatment for at least 2 weeks Consumption of a psychoactive substance - other than nicotine - within the 12 hours preceding the assessment, Presenting a score on the HAD questionnaire ≥ 11, Having benefited from a current or past RC program, Reporting to be pregnant or nursing, Current participation or in the past month in a pharmacological research protocol, Presenting difficulties for the reading or writing of the French language, Being under guardianship, Presenting disorders of higher functions

* For volunteers:

Suffering from past or current pathological gambling (DSM-5 diagnosis), Having psychiatric and addictive disorders (mood disorders, anxiety disorders and disorders linked to the use of non-nicotine substance present and not stabilized, life-long psychotic syndrome, diagnosed by the MINI), endocrine or neurological disorders (Cranial trauma, neurodegenerative diseases, unbalanced epilepsy, mental retardation, etc.), Taking a non-stabilized psychotropic treatment for at least 2 weeks, Declaring to have consumed a psychoactive substance - other than nicotine - within the 12 hours preceding the assessment, Presenting a score on the HAD questionnaire ≥ 11, Having benefited from an assumption in current or past RC program, Reporting to be pregnant or nursing, Currently participating or in the past month to a pharmacological research protocol, Presenting difficulties for the reading or writing of the French language, Being under guardianship, Presenting disorders of cognitive functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Mean difference of the scores obtained at the various neurocognitive tests between the group of disordered gamblers and the group of healthy controls | 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL BRONNEC, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hurel E, Grall-Bronnec M, Thiabaud E, Saillard A, Hardouin JB, Challet-Bouju G. A Case-Control Study on Behavioral Addictions and Neurocognition: Description of the BANCO and BANCO2 Protocols. Neuropsychiatr Dis Treat. 2021 Jul 20;17:2369-2386. doi: 10.2147/NDT.S292490. eCollection 2021. PMID 34321880